CLINICAL TRIAL: NCT04065828
Title: Oral Status and Care Needs of People Aged 90 and Over in Gironde and Dordogne
Brief Title: Oral Status and Care Needs of People Aged 90 and Over
Acronym: PAQUIDENT25
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2013/04
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Oral Health; Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will help describe the state of oral health of very old people (over 90).

DETAILED DESCRIPTION:
In 2011, according to the French National Institute for Statistics and Economic Research, people aged 85 and over accounted for about 3% of the total population. This proportion will increase sharply due to longer life expectancy on the baby boom generation and is expected to reach 7.5% of the total population in 2050.

This very old population has specific health, related to the presence of co-morbidities and co-medications, but also to a frequent state of dependence.

These general health problems and their treatment can create or accentuate oral problems or complicate their management. Thus, very old people are more likely to have some oral diseases although there is no epidemiological data in France. Conversely, oral problems can have repercussions in terms of quality of life, social relations and nutrition, and are factors of risk or aggravating actual or potential systemic disorders.

This very elderly population is therefore likely to present new challenges of dental care that it is important to document.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 90 years old
* Follow-up in 2013-2014 as part of the PAQUID cohort
* Participation Agreement

Exclusion Criteria:

* Inability to give informed consent and refusal of legal guardian.

Ages: 90 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is an ancillary study of the PAQUID cohort, of a cross-sectional nature, descriptive in a representative sample of very elderly people (≥90 years) in the Gironde and Dordogne, monocentric, with home collection.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

PRIMARY OUTCOMES:
State of the mouth and teeth | Inclusion visit
  Number of decayed, absent and closed teeth
Masticatory ability | Inclusion visit
  Number of functional units
Root caries index | Inclusion visit
  Root caries index (RCI) - RCI is based on the requirement that gingival recession must occur before root caries surface lesion begin, therefore only teeth with gum recession are examined.
  * 4 surfaces of root are examined (mesial, distal, lingual, and buccal or labial)
  * A judgment of no gum recession is made if CEJ (cement enamel junction) cannot be visualized.
  The root caries index is calculated for an individual using the formula
  • RCI= (R-D) +(R-F) x 100 (R-D) +(R-F) +(R-N) R-N =Recession present surface normal or sound R-D =Recession present with decay root surface R-F= Recession present with a filled root surface.
Hygiene index | Inclusion visit
  Hygiene index (OHI-S, Simplified Oral Hygiene Index ; from 0 to 3)
Oral pain | Inclusion visit
  Presence of oral pain yes/no
Oral lesions | Inclusion visit
  Presence and nature of oral lesions according to the International Classification of Diseases applied to odontology and stomatology of the World Health Organization
Hyposalivation / xerostomia | Inclusion visit
  Presence of hyposalivation / xerostomia (Xerostomia Inventory, XI, 11 items questionary)

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARRIVE, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khoury C, Samot J, Helmer C, Rosa RW, Georget A, Dartigues JF, Arrive E. The association between oral health and nutritional status in older adults: a cross-sectional study. BMC Geriatr. 2022 Jun 10;22(1):499. doi: 10.1186/s12877-022-03133-0. PMID 35689206
- [Derived] Rosa RW, Samot J, Helmer C, Pourtau G, Dupuis V, Fricain JC, Georget A, Dartigues JF, Arrive E. Important oral care needs of older French people: A cross-sectional study. Rev Epidemiol Sante Publique. 2020 Apr;68(2):83-90. doi: 10.1016/j.respe.2020.01.135. Epub 2020 Feb 25. PMID 32111348